CLINICAL TRIAL: NCT07267676
Title: Comparative Effects of Different Music Genres on Anxiety in Orthodontic Patients: A Randomized Controlled Study
Brief Title: Different Music Genres on Anxiety in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Alaattin Tekeli, Assist. Prof., Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025/10
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-06

CONDITIONS: Orthodontic Appliance
Keywords: Orthodontics; Music Therapy; Turkish Classical Music; Dental Anxiety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): Turkish classical music group
  Interventions: Behavioral: Turkish classical music
- Group II (Active Comparator): Patient selected music group
  Interventions: Behavioral: Patient selected music
- Group III (No Intervention): Silence

INTERVENTIONS:
Behavioral: Patient selected music — Patient selected music
  Arms: Group II
Behavioral: Turkish classical music — Patients will listen to Turkish classical music
  Arms: Group I

SUMMARY:
The goal of this clinical trial is to learn if Turkish classical music, patient-selected music, and silence have an effect on psychological and physiological anxiety indicators during orthodontic bracket placement. The main questions it aims to answer are: Does Turkish classical music reduce anxiety levels in orthodontic patients undergoing bracket placement? Does patient-selected music reduce anxiety levels in orthodontic patients undergoing bracket placement? Researchers will compare two different music genres to a control (no music, silence) to see if music therapy works to lower anxiety. Participants will: Listen to Turkish classical music or patient-selected music or silence during orthodontic bracket application and complete 2 scales before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have completed informed consent and written consent forms
* Patients between the ages of 12-18
* Patients that were undergoing orthodontic treatment and scheduled for placement of bracket appliance.

Exclusion Criteria:

* Patients over the age of 18 and below the age of 12 years
* Patients with significant medical history (psychological disorders as anxiety or depression, hearing problems, epilepsy, attention disorders, diabetes, hypertension or other systemic chronic or endocrine diseases)
* Patients using;
* psychiatric medications
* antihistaminic
* anticholinergic drugs
* Patients that did not desire to continue or participate in the research

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Levels Measured by the Abeer Children Dental Anxiety Scale (ACDAS) | Baseline (before bracket placement) and immediately after bracket placement (within 30 minutes after the intervention)
  The Abeer Children Dental Anxiety Scale (ACDAS) measures dental anxiety in children and adolescents. Scores range from 13 to 39, with higher scores indicating higher anxiety.
Change in State Anxiety Measured by the State-Trait Anxiety Inventory - State Form (STAI-S) | Baseline (before bracket placement) and immediately after bracket placement (within 30 minutes after the intervention)
  The State-Trait Anxiety Inventory State Form (STAI-S) assesses temporary state anxiety levels. Scores range from 20 to 80, with higher scores indicating higher anxiety.
Physiological Anxiety Indicators (Heart Rate, Blood Pressure, Body Temperature, Oxygen Saturation) | Baseline (before bracket placement) and immediately after bracket placement (within 30 minutes after the intervention)
  Changes in heart rate (beats per minute), blood pressure (mmHg), body temperature (degrees celcius) and oxygen saturation (%) will be recorded as indicators of physiological anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No